CLINICAL TRIAL: NCT06207591
Title: Investigation on the Cortical Communication (CortiCom) System
Brief Title: Investigation on the Cortical Communication System
Acronym: CortiCom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Erik Aarnoutse, PhD, Study Coordinator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCU 23-171; NL81205.041.23 (Other: NedMec)
Record Dates: First submitted 2023-12-01; First posted 2024-01-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Locked-in Syndrome; Neuromuscular Diseases; Brainstem Stroke; Traumatic Brain Injury
Keywords: Locked-in; Amyotrophic lateral sclerosis; Neurodegenerative disease
MeSH Terms: conditions — Locked-In Syndrome; Neuromuscular Diseases; Brain Stem Infarctions; Brain Injuries, Traumatic; Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases | interventions — Electrocorticography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECoG (electrocorticography) sensing (Experimental): Use implantable ECoG-based Brain Computer interface to control assistive technology
  Interventions: Device: ECoG (electrocorticography) sensing

INTERVENTIONS:
Device: ECoG (electrocorticography) sensing — Implant electrodes and pedestal connector and use, through amplifier and decoding, for control of BCI
  Other Names: CortiCom-Utrecht assembly

SUMMARY:
The goal of this clinical trial is to demonstrate communication through a brain implant in people in locked-in state, i.e. people with severe paralysis and communication problems.

The main questions it aims to answer are efficient and stable control of Brain-Computer interface (BCI) functions for communication with attempted hand movements and operation of a keyword-based speech BCI.

Participants will be implanted with four electrode grids, with in total 128 electrodes, on the surface of the brain and a connector on the skull. Participation includes visits of researchers for recording and training at home, 2-3 times per week for one year. Extension of participation after one year is possible.

If successful, the participant will be able to use the BCI at home independently, without the presence of a researcher.

DETAILED DESCRIPTION:
Locked-In Syndrome (LIS) is a neurological condition in which communication is impossible, or profoundly impaired, due to loss of speech and other motor functions, while cognition is intact. The most distressing aspect of LIS is the inability to initiate and sustain communication. Existing assistive technologies (ATs) fall short of a remedy. An effective brain-computer interface (BCI) for communication would dramatically improve quality of life for people with LIS. Electrocorticography (ECoG) with non-penetrating subdural electrodes is a promising implantable approach for BCI. In this study, the "CortiCom system" (which stands for Cortical Communication) wil be used. This system combines an implantable assembly, consisting of four small high-density (HD) ECoG grids on the hand and speech areas of the motor cortex, totalling 128-channels, and a transcutaneous pedestal connector, with an external data acquisition system. With the CortiCom system the overall hypothesis will be tested that broader and more densely spaced ECoG electrodes can better tap into the spatial detail of the organization of the sensorimotor cortex in order to expand BCI function and restore meaningful communication in LIS. Specifically, the CortiCom system will substantially increase the number and density of electrodes recording from the brain to determine whether more sophisticated control and communication can be achieved with more comprehensive and detailed spatial sampling of representations for movements of the hand/arm and of speech articulators. Clinically meaningful outcomes for people with LIS include rapid reestablishment, and stable maintenance of communication, at minimum consisting of a caregiver call-button and menu selections.

Objective:

Primary Objective 1: Demonstrate efficient and stable control of essential BCI functions (initiate BCI, call caregiver, and menu selections). Primary Objective 2: Demonstrate efficient and stable operation of a keyword-based speech BCI.

Intervention:

Participants will be implanted with an assembly consisting of HD-ECoG electrode grids over the sensorimotor cortex and a transcutaneous pedestal connector. The assembly will be connected with an external data acquisition system during recordings. During recordings, feedback about the neural signals is given via a visual display and participants are trained to employ the neural signals for fast brain-based communication. Upon adequate performance, participants can independently (i.e., without researcher involvement) train with and use the system at home for validation of performance and usability. After implantation, participation has a duration of 1 year, with a possibility of extension.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* Clinical diagnosis of locked-in state state or likelihood of soon progressing into LIS (within an estimated 2 years), caused by traumatic brain injury, brainstem stroke, neurodegenerative disease, neuromuscular disease or another cause
* • Current or imminent complete or incomplete tetraplegia (quadriplegia) or tetraparesis (quadriparesis)
* • Current or imminent motor-related speech impairment (dysarthria or anarthria)
* Either receiving tracheostomy invasive ventilation, or having a stable and adequate respiratory situation without respiratory support, allowing for safe intubation, mechanical ventilation and detubation during surgery according to the involved clinicians, and, if relevant (e.g., in case of a progressive condition), in combination with a confirmed desire to receive tracheostomy invasive ventilation when that becomes necessary
* Meeting surgical safety criteria, including surgical clearance by the study physicians
* Meeting (neuro)psychological evaluation criteria
* Ability to communicate reliably, such as through eye movement
* Willingness and ability to provide informed consent
* Lives within reasonable distance from University Medical Center Utrecht
* Participant consents to the study and still wishes to participate at the time of the study
* Vision and hearing largely intact

Exclusion Criteria:

* Performance on formal neuropsychological testing that indicates a significant current or recent psychiatric disorder, cognitive or behavioral impairment, that would interfere with obtaining informed consent or fully participating in study activities
* Medical conditions contraindicating surgery of a chronically implanted device or that could interfere with study participation (for example active infections, unexplained fever, existing scalp lesions or skin breakdown, osteomyelitis, hepatitis, any autoimmune disease/disorder, epilepsy, skin disorders causing excessive skin sloughing or poor wound healing, cranioplasty, significant cardiovascular, metabolic, or renal impairments, chronic oral or intravenous use of steroids or immunosuppressive therapy, active cancer within the past year or requires chemotherapy, uncontrolled autonomic dysreflexia within the past 3 months, hydrocephalus with or without an implanted ventricular shunt or a medical contraindication to stop anti-coagulant medications during surgery)
* Presence of pre-surgical findings in anatomical, functional, and/or vascular neuroimaging that makes achieving implant locations too challenging or incompatible with desired risk levels
* Inability to undergo MRI for pre-implantation evaluation, for example due to the presence of implanted devices that are incompatible with MRI, which may include pacemakers, cardiac defibrillators, spinal cord or vagal nerve stimulators, deep brain stimulators, and cochlear implants
* Anticipated need for MRI after implantation of the CortiCom assembly

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Usability of the BCI system - Accuracy | 1 year
  Accuracy: >80% sensitivity (true positive rate) for 1-command control, and 90% sensitivity and 80% classification accuracy (distinguishing between the six classes) for 6-command control
Usability of the BCI system - speed | 1 year
  Speed characters or keywords per minute
Usability of the BCI system - subjective workload Visual Analogue Scale (VAS) | 1 year
  Subjective Workload: Visual Analogue Scale Continuous scale: Little to no effort (0) - Much effort (5). Lower numbers are better.
Usability of the BCI system - subjective workload National Aeronautics and Space Administration-Task Load Index (NASA-TLX) | 1 year
  Subjective Workload: National Aeronautics and Space Administration-Task Load Index Scale: 21 point Likert-type scale. Lower numbers are better.
Usability of the BCI system - user satisfaction Psychosocial impact of assistive devices scale (PIADS) | 1 year
  User Satisfaction: Psychosocial impact of assistive devices scale. Likert-type scale -3, -2, -1, 0, 1, 2, 3. 3 is best result.
Usability of the BCI system - user satisfaction Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) | 1 year
  User Satisfaction: Quebec User Evaluation of Satisfaction with assistive Technology version 2.0.
  Likert-type scale: Extremely dissatisfied - Dissatisfied - Slightly satisfied - Satisfied - Extremely satisfied. Extremely Satisfied is the best result.
Usability of the BCI system - validation | 1 year
  Validation: Questionnaire to evaluate user satisfaction and ease of use of the home use software.
  Likert-type scale: fully disagree - disagree - neither agree or disagree - agree - fully agree - not applicable. Fully agree is the best result.
Degrees of Freedom of BCI Control. | 1 year
  the number of different commands that are successfully decoded, or the size of the decoded vocabulary

SECONDARY OUTCOMES:
Stability of BCI performance (electrode-tissue interaction) | 2 years
  Longitudinal data of the 24-hour cycle after implantation of the impedance (in Ω). The data are fitted to determine trends and variance, over weeks, to determine improvement or deterioration of electrode-tissue interaction.
Stability of BCI performance (signal) | 2 years
  Longitudinal data of the 24-hour cycle after implantation of the raw power (after wavelet transform, in arbitrary units). The data are fitted to determine trends and variance, both within 24 hrs to detect a possible circadian pattern and over weeks, to determine improvement or deterioration of signal amplitude.
Stability of BCI performance (modulation) | 2 years
  Longitudinal data of the 24-hour cycle after implantation of the task-related modulation in power (correlation in r2). The data are fitted to determine trends and variance, over weeks, to determine improvement or deterioration of modulation.
Stability of BCI performance (performance) | 2 years
  Longitudinal data of the 24-hour cycle after implantation of the BCI performance (task accuracy). The data are fitted to determine trends and variance, both within 24 hrs to detect a possible circadian pattern and over weeks, to see improvement or deterioration of accuracy.
Independent use of BCI | 2 years
  Longitudinal data of independent use per day. The best result is 24h use. The data are fitted to determine trends and variance, both within 24 hrs to detect a possible circadian pattern and over weeks, to see increase or decrease of the hours of independent use.

OTHER OUTCOMES:
Assess device specifications for future application of HD ECoG-BCIs | 2 years
  qualitative description on device specifications and experimental parameters, such as the specific decoder settings, for future, larger scale, application of HD ECoG-BCIs.

CONTACTS AND LOCATIONS:
Overall Officials: Nick F Ramsey, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
selected datasets will be available through a public repository after publication of results
Time Frame: after first published results, no end date
Access Criteria: Publicly available

REFERENCES:
- [Background] Vansteensel MJ, Leinders S, Branco MP, Crone NE, Denison T, Freudenburg ZV, Geukes SH, Gosselaar PH, Raemaekers M, Schippers A, Verberne M, Aarnoutse EJ, Ramsey NF. Longevity of a Brain-Computer Interface for Amyotrophic Lateral Sclerosis. N Engl J Med. 2024 Aug 15;391(7):619-626. doi: 10.1056/NEJMoa2314598. PMID 39141854
- [Background] Vansteensel MJ, Pels EGM, Bleichner MG, Branco MP, Denison T, Freudenburg ZV, Gosselaar P, Leinders S, Ottens TH, Van Den Boom MA, Van Rijen PC, Aarnoutse EJ, Ramsey NF. Fully Implanted Brain-Computer Interface in a Locked-In Patient with ALS. N Engl J Med. 2016 Nov 24;375(21):2060-2066. doi: 10.1056/NEJMoa1608085. Epub 2016 Nov 12. PMID 27959736
- [Result] The neural representation of fine hand movements in an individual approaching locked-in syndrome (2025) S.H. Geukes, A. Bekius, M.P. Branco, M.S.W. Verberne, A. Schippers, Z.V. Freudenburg, E.J. Aarnoutse, M.J. Vansteensel, N.E. Crone, N.F. Ramsey. 11th International BCI Meeting, Banff, Canada, DOI: 10.3217/978-3-99161-050-2-085